CLINICAL TRIAL: NCT01149590
Title: Role of Multidetector Computed Tomography in the Diagnosis and Management of Patients Attending a Rapid Access Chest Pain Clinic
Brief Title: Scottish COmputed Tomography of the HEART Trial
Acronym: SCOT-HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CZH/4/588
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2017-04

CONDITIONS: Angina Pectoris; Coronary Heart Disease
Keywords: Angina; Coronary Heart Disease; Computed Tomography; Angiogram; Coronary Artery Calcium Score; Chest Pain; Angina Pectoris due to Coronary Heart Disease
MeSH Terms: conditions — Angina Pectoris; Coronary Disease; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT Calcium Score & Coronary Angiography (Experimental): CT Scan
  Interventions: Procedure: Computer Tomography Angiography
- No CT Scan (No Intervention): No CT Scan

INTERVENTIONS:
Procedure: Computer Tomography Angiography — Computed Tomography Angiography
  Arms: CT Calcium Score & Coronary Angiography

SUMMARY:
The primary objective of the study is to see if coronary artery calcium score and computed tomography coronary angiogram alters the proportion of patients diagnosed with angina due to coronary heart disease.

DETAILED DESCRIPTION:
Rapid access chest pain clinics have facilitated the early diagnosis and treatment of patients with coronary heart disease and angina. Despite this important service provision, coronary heart disease continues to be under-diagnosed and many patients are left untreated and at risk. Recent advances in imaging technology have now led to the widespread use of non-invasive computed tomography both to measure coronary artery calcium scores and undertake coronary angiography. However, this technology has not been robustly evaluated in any systematic approach. Using state-of-the-art multidetector computed tomography scanners, we propose to undertake a major multicentre randomized controlled trial to assess the added value of computed tomography imaging in over 4000 patients attending rapid access chest pain clinics across Scotland. This will define the most appropriate use of this emerging technology in the setting of diagnosing and treating patients with coronary heart disease and angina pectoris. This study will also lay the foundation for future studies to look at the potential prognostic value of this technology.

ELIGIBILITY:
Inclusion Criteria:

* 18 and ≤75 years of age
* Attendance at the Rapid Access Chest Pain Clinic

Exclusion Criteria:

* Inability or unwilling to undergo computed tomography scanning, such as exceeding weight tolerance of scanner
* Severe renal failure (serum creatinine >200 µmol/L or estimated glomerular filtration rate <30 mL/min)
* Previous recruitment to the trial
* Major allergy to iodinated contrast agent
* Unable to give informed consent
* Known pregnancy
* Acute coronary syndrome within 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4138 (Actual)
Dates: Start 2010-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with angina pectoris secondary to coronary heart disease | 6 weeks

SECONDARY OUTCOMES:
Symptoms | Baseline, after computed tomography scan (where appropriate), 6 weeks and 6 months
  (i) Chest pain. (ii) Quality of life.
Diagnosis | Baseline, after computed tomography scan (where appropriate), 6 weeks and 6 months
  (i) Diagnosis and severity of coronary heart disease (ii) Accuracy of computed tomography coronary angiography
Investigations | Baseline, 6 weeks, 6 months
  (i) Exercise electrocardiographic stress test (ii) Nuclear medicine imaging - myocardial perfusion imaging (iii) Stress echocardiography (iv) Invasive coronary angiography (v) Non-coronary investigations
Treatment | Baseline, after computed tomography scan (where appropriate), 6 weeks, 6 months
  (i) Secondary prevention (ii) Pharmacological anti-anginal therapy (iii) Coronary revascularisation
Long-term outcome | 10 years
  (i) Coronary heart disease death or non-fatal Myocardial Infarction (MI) (ii) Coronary heart disease death (iii) Non-fatal MI (iv) Coronary heart disease death, non-fatal MI or non-fatal stroke (v) Non-fatal stroke (vi) All-cause death (vii) Cardiovascular death (viii) Coronary revascularisation; percutaneous coronary intervention or coronary artery bypass graft surgery (ix) Hospitalisation for chest pain including acute coronary syndromes and non-coronary chest pain (x) Hospitalisation for cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral arterial disease

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, BA BSc BM DM PhD FRCP DSc, Principal Investigator — University of Edinburgh
Locations (12):
- United Kingdom (12):
  - Borders General Hospital, Melrose, Borders
  - Victoria Hospital, Kirkcaldy, Fife
  - Ninewells Hospital, Dundee, Tayside
  - University Hospital Ayr, Ayr
  - Royal Infirmary Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh
  - Western Infirmary Glasgow, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Forth Valley Royal, Larbert
  - St John's Hosptial, Livingston
  - Royal Alexandra Hospital, Paisley
  - Perth Royal Infirmary, Perth

IPD SHARING:
Plan to Share IPD: Yes
Please contact corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: Post primary publication

REFERENCES:
- [Background] Newby DE, Williams MC, Flapan AD, Forbes JF, Hargreaves AD, Leslie SJ, Lewis SC, McKillop G, McLean S, Reid JH, Sprat JC, Uren NG, van Beek EJ, Boon NA, Clark L, Craig P, Flather MD, McCormack C, Roditi G, Timmis AD, Krishan A, Donaldson G, Fotheringham M, Hall FJ, Neary P, Cram L, Perkins S, Taylor F, Eteiba H, Rae AP, Robb K, Barrie D, Bissett K, Dawson A, Dundas S, Fogarty Y, Ramkumar PG, Houston GJ, Letham D, O'Neill L, Pringle SD, Ritchie V, Sudarshan T, Weir-McCall J, Cormack A, Findlay IN, Hood S, Murphy C, Peat E, Allen B, Baird A, Bertram D, Brian D, Cowan A, Cruden NL, Dweck MR, Flint L, Fyfe S, Keanie C, MacGillivray TJ, Maclachlan DS, MacLeod M, Mirsadraee S, Morrison A, Mills NL, Minns FC, Phillips A, Queripel LJ, Weir NW, Bett F, Divers F, Fairley K, Jacob AJ, Keegan E, White T, Gemmill J, Henry M, McGowan J, Dinnel L, Francis CM, Sandeman D, Yerramasu A, Berry C, Boylan H, Brown A, Duffy K, Frood A, Johnstone J, Lanaghan K, MacDuff R, MacLeod M, McGlynn D, McMillan N, Murdoch L, Noble C, Paterson V, Steedman T, Tzemos N. Role of multidetector computed tomography in the diagnosis and management of patients attending the rapid access chest pain clinic, The Scottish computed tomography of the heart (SCOT-HEART) trial: study protocol for randomized controlled trial. Trials. 2012 Oct 4;13:184. doi: 10.1186/1745-6215-13-184. PMID 23036114
- [Result] SCOT-HEART investigators. CT coronary angiography in patients with suspected angina due to coronary heart disease (SCOT-HEART): an open-label, parallel-group, multicentre trial. Lancet. 2015 Jun 13;385(9985):2383-91. doi: 10.1016/S0140-6736(15)60291-4. Epub 2015 Mar 15. PMID 25788230
- [Result] SCOT-HEART Investigators; Newby DE, Adamson PD, Berry C, Boon NA, Dweck MR, Flather M, Forbes J, Hunter A, Lewis S, MacLean S, Mills NL, Norrie J, Roditi G, Shah ASV, Timmis AD, van Beek EJR, Williams MC. Coronary CT Angiography and 5-Year Risk of Myocardial Infarction. N Engl J Med. 2018 Sep 6;379(10):924-933. doi: 10.1056/NEJMoa1805971. Epub 2018 Aug 25. PMID 30145934
- [Derived] Rasmussen LD, Sikjaer M, Soby JH, Pedersen OB, Westra J, Efthekhari A, Christiansen EH, Foldyna B, Williams MC, Dweck MR, Newby DE, Douglas PS, Bottcher M, Winther S. Dual probability approach for risk adjustment in patients with a low clinical likelihood of coronary artery disease. Eur Heart J Cardiovasc Imaging. 2025 Aug 29;26(9):1507-1517. doi: 10.1093/ehjci/jeaf193. PMID 40590244
- [Derived] Williams MC, Wereski R, Tuck C, Adamson PD, Shah ASV, van Beek EJR, Roditi G, Berry C, Boon N, Flather M, Lewis S, Norrie J, Timmis AD, Mills NL, Dweck MR, Newby DE; SCOT-HEART Investigators. Coronary CT angiography-guided management of patients with stable chest pain: 10-year outcomes from the SCOT-HEART randomised controlled trial in Scotland. Lancet. 2025 Jan 25;405(10475):329-337. doi: 10.1016/S0140-6736(24)02679-5. PMID 39863372
- [Derived] Kolossvary M, Lin A, Kwiecinski J, Cadet S, Slomka PJ, Newby DE, Dweck MR, Williams MC, Dey D. Coronary Plaque Radiomic Phenotypes Predict Fatal or Nonfatal Myocardial Infarction: Analysis of the SCOT-HEART Trial. JACC Cardiovasc Imaging. 2025 Mar;18(3):308-319. doi: 10.1016/j.jcmg.2024.08.012. Epub 2024 Oct 30. PMID 39480364
- [Derived] Williams MC, Kwiecinski J, Doris M, McElhinney P, D'Souza MS, Cadet S, Adamson PD, Moss AJ, Alam S, Hunter A, Shah ASV, Mills NL, Pawade T, Wang C, Weir-McCall JR, Bonnici-Mallia M, Murrills C, Roditi G, van Beek EJR, Shaw LJ, Nicol ED, Berman DS, Slomka PJ, Newby DE, Dweck MR, Dey D. Sex-Specific Computed Tomography Coronary Plaque Characterization and Risk of Myocardial Infarction. JACC Cardiovasc Imaging. 2021 Sep;14(9):1804-1814. doi: 10.1016/j.jcmg.2021.03.004. Epub 2021 Apr 14. PMID 33865779
- [Derived] Singh T, Bing R, Dweck MR, van Beek EJR, Mills NL, Williams MC, Villines TC, Newby DE, Adamson PD. Exercise Electrocardiography and Computed Tomography Coronary Angiography for Patients With Suspected Stable Angina Pectoris: A Post Hoc Analysis of the Randomized SCOT-HEART Trial. JAMA Cardiol. 2020 Aug 1;5(8):920-928. doi: 10.1001/jamacardio.2020.1567. PMID 32492104
- [Derived] Williams MC, Kwiecinski J, Doris M, McElhinney P, D'Souza MS, Cadet S, Adamson PD, Moss AJ, Alam S, Hunter A, Shah ASV, Mills NL, Pawade T, Wang C, Weir McCall J, Bonnici-Mallia M, Murrills C, Roditi G, van Beek EJR, Shaw LJ, Nicol ED, Berman DS, Slomka PJ, Newby DE, Dweck MR, Dey D. Low-Attenuation Noncalcified Plaque on Coronary Computed Tomography Angiography Predicts Myocardial Infarction: Results From the Multicenter SCOT-HEART Trial (Scottish Computed Tomography of the HEART). Circulation. 2020 May 5;141(18):1452-1462. doi: 10.1161/CIRCULATIONAHA.119.044720. Epub 2020 Mar 16. PMID 32174130
- [Derived] Adamson PD, Williams MC, Dweck MR, Mills NL, Boon NA, Daghem M, Bing R, Moss AJ, Mangion K, Flather M, Forbes J, Hunter A, Norrie J, Shah ASV, Timmis AD, van Beek EJR, Ahmadi AA, Leipsic J, Narula J, Newby DE, Roditi G, McAllister DA, Berry C; SCOT-HEART Investigators. Guiding Therapy by Coronary CT Angiography Improves Outcomes in Patients With Stable Chest Pain. J Am Coll Cardiol. 2019 Oct 22;74(16):2058-2070. doi: 10.1016/j.jacc.2019.07.085. PMID 31623764
- [Derived] Bing R, Henderson J, Hunter A, Williams MC, Moss AJ, Shah ASV, McAllister DA, Dweck MR, Newby DE, Mills NL, Adamson PD. Clinical determinants of plasma cardiac biomarkers in patients with stable chest pain. Heart. 2019 Nov;105(22):1748-1754. doi: 10.1136/heartjnl-2019-314892. Epub 2019 Jun 1. PMID 31154425
- [Derived] Williams MC, Moss AJ, Dweck M, Adamson PD, Alam S, Hunter A, Shah ASV, Pawade T, Weir-McCall JR, Roditi G, van Beek EJR, Newby DE, Nicol ED. Coronary Artery Plaque Characteristics Associated With Adverse Outcomes in the SCOT-HEART Study. J Am Coll Cardiol. 2019 Jan 29;73(3):291-301. doi: 10.1016/j.jacc.2018.10.066. PMID 30678759
- [Derived] Adamson PD, Hunter A, Madsen DM, Shah ASV, McAllister DA, Pawade TA, Williams MC, Berry C, Boon NA, Flather M, Forbes J, McLean S, Roditi G, Timmis AD, van Beek EJR, Dweck MR, Mickley H, Mills NL, Newby DE. High-Sensitivity Cardiac Troponin I and the Diagnosis of Coronary Artery Disease in Patients With Suspected Angina Pectoris. Circ Cardiovasc Qual Outcomes. 2018 Feb;11(2):e004227. doi: 10.1161/CIRCOUTCOMES.117.004227. PMID 29444926
- [Derived] Adamson PD, Fordyce CB, McAllister DA, Udelson JE, Douglas PS, Newby DE. Identification of patients with stable chest pain deriving minimal value from coronary computed tomography angiography: An external validation of the PROMISE minimal-risk tool. Int J Cardiol. 2018 Feb 1;252:31-34. doi: 10.1016/j.ijcard.2017.09.033. PMID 29249436
- [Derived] Adamson PD, Hunter A, Williams MC, Shah ASV, McAllister DA, Pawade TA, Dweck MR, Mills NL, Berry C, Boon NA, Clark E, Flather M, Forbes J, McLean S, Roditi G, van Beek EJR, Timmis AD, Newby DE. Diagnostic and prognostic benefits of computed tomography coronary angiography using the 2016 National Institute for Health and Care Excellence guidance within a randomised trial. Heart. 2018 Feb;104(3):207-214. doi: 10.1136/heartjnl-2017-311508. Epub 2017 Aug 27. PMID 28844992
- [Derived] McCarter RV, McKay GJ, Quinn NB, Chakravarthy U, MacGillivray TJ, Robertson G, Pellegrini E, Trucco E, Williams MC, Peto T, Dhillon B, van Beek EJ, Newby DE, Kee F, Young IS, Hogg RE. Evaluation of coronary artery disease as a risk factor for reticular pseudodrusen. Br J Ophthalmol. 2018 Apr;102(4):483-489. doi: 10.1136/bjophthalmol-2017-310526. Epub 2017 Aug 19. PMID 28822985
- [Derived] Williams MC, Hunter A, Shah A, Assi V, Lewis S, Mangion K, Berry C, Boon NA, Clark E, Flather M, Forbes J, McLean S, Roditi G, van Beek EJ, Timmis AD, Newby DE; Scottish COmputed Tomography of the HEART (SCOT-HEART) Trial Investigators. Symptoms and quality of life in patients with suspected angina undergoing CT coronary angiography: a randomised controlled trial. Heart. 2017 Jul;103(13):995-1001. doi: 10.1136/heartjnl-2016-310129. Epub 2017 Feb 28. PMID 28246175
- [Derived] Williams MC, Hunter A, Shah ASV, Assi V, Lewis S, Smith J, Berry C, Boon NA, Clark E, Flather M, Forbes J, McLean S, Roditi G, van Beek EJR, Timmis AD, Newby DE; SCOT-HEART Investigators. Use of Coronary Computed Tomographic Angiography to Guide Management of Patients With Coronary Disease. J Am Coll Cardiol. 2016 Apr 19;67(15):1759-1768. doi: 10.1016/j.jacc.2016.02.026. PMID 27081014
- [Derived] Moss AJ, Newby DE. CT coronary angiographic evaluation of suspected anginal chest pain. Heart. 2016 Feb 15;102(4):263-8. doi: 10.1136/heartjnl-2015-307860. Epub 2015 Dec 8. PMID 26647079
- [Derived] Williams MC, Golay SK, Hunter A, Weir-McCall JR, Mlynska L, Dweck MR, Uren NG, Reid JH, Lewis SC, Berry C, van Beek EJ, Roditi G, Newby DE, Mirsadraee S. Observer variability in the assessment of CT coronary angiography and coronary artery calcium score: substudy of the Scottish COmputed Tomography of the HEART (SCOT-HEART) trial. Open Heart. 2015 May 19;2(1):e000234. doi: 10.1136/openhrt-2014-000234. eCollection 2015. PMID 26019881